CLINICAL TRIAL: NCT03308279
Title: Ultrasound and Anthropometric Prediction Model for Minimizing the Risk of Median Nerve Puncture With Dry Needling Approach Into the Pronator Teres Muscle
Brief Title: Prediction Model for Minimizing the Risk of Median Nerve Puncture
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Prof. Raúl Ferrer Peña, Universidad Autonoma de Madrid
Other Study IDs: Pronator Teres Prediction
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Pronator Teres Nerve Syndrome
Keywords: dry needling; median nerve; Pronator Teres
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asinthomatic: The only group evaluated
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound and Anthropometric meassures
  Other Names: Anthropometric meassures

SUMMARY:
The main aim of this study was to correlate anthropometric measures of the forearm in healthy subjects with the ultrasound pronator teres depth to determine the needle length in order to avoid injury of the median nerve during pronator teres dry needle approach. A cross-sectional study, was carried out in order to perform a predictive model for the median nerve depth into the pronator teres muscle using a decision tree analysis algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Asinthomatic subjets

Exclusion Criteria:

* Pain in the 3 moths before in the forearm

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asinthomatic subjets who respond to the researchers calls
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Muscle thicknesses | 10 minutes
  With ultrasound
Median Nerve depth | 5 minutes
  With ultrasound
Forearm Perimeter | 2 minutes
  in cm
Forearm Longitude | 2 minutes
  in cm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurses IA, Altinel L, Gayretli O, Akgul T, Uzun I, Dikici F. Morphology and morphometry of the ulnar head of the pronator teres muscle in relation to median nerve compression at the proximal forearm. Orthop Traumatol Surg Res. 2016 Dec;102(8):1005-1008. doi: 10.1016/j.otsr.2016.08.016. Epub 2016 Nov 11. PMID 27843079
- [Background] Dang AC, Rodner CM. Unusual compression neuropathies of the forearm, part II: median nerve. J Hand Surg Am. 2009 Dec;34(10):1915-20. doi: 10.1016/j.jhsa.2009.10.017. PMID 19969200
- [Background] Kowalska B, Sudol-Szopinska I. Ultrasound assessment on selected peripheral nerve pathologies. Part I: Entrapment neuropathies of the upper limb - excluding carpal tunnel syndrome. J Ultrason. 2012 Sep;12(50):307-18. doi: 10.15557/JoU.2012.0016. Epub 2012 Sep 30. PMID 26674101